CLINICAL TRIAL: NCT00888394
Title: Clinical Effectiveness of Quiropodiatry and Orthesis on Heel and Plantar Pain: Randomized Control Trial
Brief Title: Effectiveness of Podiatry on Plantar Pain
Acronym: EPOPLAPAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 173908909-8909-4-9
Record Dates: First submitted 2009-04-22; First posted 2009-04-27 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-01

CONDITIONS: Heel Pain; Plantar Fasciitis; Plantar Pain
Keywords: chiropody; podiatry; insoles; foot orthesis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Procedure: chiropody
- 2 (Experimental)
  Interventions: Procedure: basic orthesis
- 3 (Experimental)
  Interventions: Procedure: advantage orthesis
- 4 (Experimental)
  Interventions: Procedure: chiropody and advantage orthesis

INTERVENTIONS:
Procedure: chiropody — basic procedure of chiropody in podiatry
  Arms: 1
Procedure: basic orthesis — individual basic orthesis of foot
  Arms: 2
Procedure: advantage orthesis — advantage orthesis of foot with special material and design
  Arms: 3
Procedure: chiropody and advantage orthesis — chiropody and advantage orthesis of foot
  Arms: 4

SUMMARY:
MAIN OBJECTIVE: To value the effectiveness of the different quiropody interventions in the heel pain.

SECONDARY OBJECTIVES: To evaluate the effectiveness of lasw different technologies in front of each one of the other experimental technologies. To analyze the state of general health and of quality of the patients' life in all the treatment groups. To analyze the study cost-effectiveness of each one of the experimental interventions. DESIGN: randomized controled trial, prospective.

SUBJECT OF STUDY: Patient that go to the Assistance Educational Unit of Podología of the E.U. Sciences of the Health with footpain like consultation reason.

INTERVENTION: Establishment of four experimental groups with intervention varied podológica. He/she will be carried out a complete pursuit with valuations at the 1,2, 6, 12 and 24 months, by means of pain scales and function of the foot (FHSQ), the index postural of the foot (FPI), the study of pressures by means of biofoot/IBV and of the state of general health (SF-12) and quality of life (Euroqol).

VARIABLES: Of intervention; treatment basic orthopodiatry, treatment advanced orthopodiatry, of treatment quiropody. Of result: pain and function of the foot (FHSQ), of the state of general health (SF12) and quality of life (Euroqol). Variables of characterization of the sample.

ANALYSIS DATA: Descriptive statistic, with measures of central tendency and dispersion of the study variables. They will be carried out statistical inferenciales between the main variables of intervention and result (square chi, t Student, ANOVA, Mann-Whitney, Wilcoxon, according to types and normality of variables). Likewise, measures of the size of the effect will settle down in the main variables of result, by means of the relative reduction of the risk, absolute risk and odds ratio, with their respective intervals of trust.

ELIGIBILITY:
Inclusion Criteria:

* Heel and plantar pain

Exclusion Criteria:

* Inflammatory infections and specific organic disease of foot

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Health state and pain of foot with FHSQ | total score, pre and post intervention and 6 and 12 months of follow up

SECONDARY OUTCOMES:
quality of life with EuroQoL 5D (Spanish Version) | scale 0-100, pre and post intervention and follow up 6 and 12 months
biomechanical parameters with Biofoot applications (instrumental systme of dinamic pressure inside shoes) | Kp in 68 sensors of plantar foot, changes pre-post intervention and 6 and 12 months of follow up

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clinica Podologia de la Universidad de malaga, Málaga, Malaga
  - Health Science School , University of Malaga, Málaga, Malaga

REFERENCES:
- See also: University of Malaga — http://www.uma.es/
- See also: Health Science School — http://www.salud.uma.es/
- See also: Ethics Comite Andalucia — http://www.juntadeandalucia.es/salud/principal/documentos.asp?pagina=ec_op1
- See also: R+D Spain — http://www.plannacionalidi.es/plan-idi-public/